CLINICAL TRIAL: NCT00796627
Title: HIF-1 Regulated Circulating Angiogenic Cell Recruitment in Burn Wound Healing
Brief Title: Hypoxia-inducible Factor-1 (HIF-1) Regulated Circulating Angiogenic Cells (CACs) Recruitment in Burn Wound Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit enough patients
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00018037
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Wound Healing; Burns
Keywords: Wound Healing; Burns; HIF-1; CAC
MeSH Terms: conditions — Burns

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Sham Comparator): Healthy volunteers with no burn wounds Volunteers donate blood that will be studied in comparison to patients who have sustained burns. The circulating "bone marrow stem cells" will be counted and compared to the levels in burn patients. Six 12 ml tubes will be taken for the study. You will not be compensated. But you will be helping to advance science if you join the study.
  Interventions: Genetic: Healthy volunteers
- Burn volunteer (Active Comparator): To recruit burn wound patients with defined clinical criteria for study. A second-degree burn of at least 10 cm2 to up to 95% BSA; age = 14-75 years; BP > 100 mm Hg systolic; heart rate < 100 beats/minute; urine output > 30 ml/hour; area of burn < 20% of BSA; body temperature = 98.5-101 degrees Fahrenheit; serum albumin > 3 mg/ml; and informed consent. We will also obtain a history regarding the presence or absence of risk factors that may affect CAC numbers: hypertension > 1 year; smoking > 2 pack-years or within the last year; diabetes mellitus; and family history of premature coronary artery disease (men < 55 and women < 65 years of age).Six 12 ml tubes will be taken at 5 time points
  Interventions: Other: Burn volunteers

INTERVENTIONS:
Genetic: Healthy volunteers — Comparison of healthy volunteers to burn wounded volunteers
  Arms: Healthy volunteers
Other: Burn volunteers — Comparison of burn wounded volunteers to healthy volunteers
  Other Names: Burn wounds
  Arms: Burn volunteer

SUMMARY:
This research is being done to increase knowledge about wound healing and different factors that may affect healing in burn patients.

DETAILED DESCRIPTION:
Burn injuries represent a major public health problem, requiring medical attention for more than one million Americans annually. Despite therapeutic advances, non-healing burn wounds and excessive scarring still result in significant long term physical and psychosocial morbidity. In this study we propose to perform clinical and research to study the role of circulating angiogenic cells (CAC) in promoting burn wound healing.

CAC's have been shown to contribute to vascularization and tissue repair in a number of animal models of tissue injury ischemia and mobilization of CACs into the peripheral blood has been demonstrated in burn wound patients.

We hypothesize that primary healing of burn wounds is dependent on repair of damaged vasculature, and that bone marrow derived stem cells, circulating angiogenic cells (CAC), play a critical role in the healing process. Furthermore we propose that the transcription factor Hypoxia Inducible Factor 1 alpha (HIF 1 alpha) through production of peptide products of its downstream target genes directs the "homing" of CAC's to the wound where they participate in healing events. The first aim of this study is to correlate mobilization of CAC's into the blood stream with the success of burn wound healing.

CAC's have been shown to contribute to vascularization and tissue repair in a number of studies. The relationship between mobilization of CAC's and burn wound healing has not been examined. In addition to surveying CAC numbers in the peripheral blood, we will assay levels of the putative mediators of CAC mobilization: Vascular Endothelial Growth Factor (VEGF), Placenta Growth Factor (PLGF), and Stromal Cell-Derived Factor (SDF-1). We hypothesize that individuals who are able to mount a large and sustained mobilization of CAC's into the peripheral blood from the bone marrow, will be more likely to heal the injured vasculature and go on to primary healing. Individuals with an inadequate mobilization of CAC's will fail to repair the damaged vasculature in the wound and proceed to necrosis and "conversion" to third degree, necrotic burn wounds.

ELIGIBILITY:
Inclusion Criteria:

Recruitment of patients at the Johns Hopkins Regional Burn Center for study will be based upon the following clinical criteria:

* Second degree scald burn of 10 cm2
* Age between 14 to 75 years
* Burn area equal or less than 95% of Burn Surface Area (BSA)
* Body temperature between 98.5 and 101 degree F
* Informed consent for enrolment into study
* Spanish speaking patients will be included when we have a Spanish consent form available.

Exclusion Criteria:

* First and third degree burn wounds
* Hemodynamic instability (SBP below 100, Heart Rate (HR) over 100, urine output less than 30 ml/hour
* Area of burn over 20% of BSA
* Hypothermia T<98.5 or Hyperthermia T>101 degree F
* Urine output less than 30 ml/hour
* Serum albumin less than 3 mg/ml.
* Subjects weighing less than 50 kg.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Harmon, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Wei X, Liu L, Marti GP, Ghanamah MS, Arshad MJ, Strom L, Spence R, Jeng J, Milner S, Harmon JW, Semenza GL. Association of increasing burn severity in mice with delayed mobilization of circulating angiogenic cells. Arch Surg. 2010 Mar;145(3):259-66. doi: 10.1001/archsurg.2009.285. PMID 20231626

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Healthy volunteers with no burn wounds
  Healthy volunteers: Comparison of healthy volunteers to burn wounded volunteers
- Burn Volunteer: Burn wounded volunteers
  Burn volunteers: Comparison of burn wounded volunteers to healthy volunteers
Period: Overall Study
Arm/Group | Healthy Volunteers | Burn Volunteer
Started | 10 | 31
Completed | 10 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Burn Volunteer | Total
Number analyzed (Participants) | 10 | 31 | 41
Age, Customized [Count of Participants; unit: Participants]
  >=14, <=75 | 10 | 31 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 24 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 24 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 31 | 41

OUTCOME MEASURES:

1. Primary Outcome: The Quantification of Circulating Angiogenic Cells in the Blood of Individuals Who Are Healthy Volunteers Compared to Those in Individuals Who Have Sustained a Burn Injury
Description: Tissue samples were harvested from healthy volunteers and participants who sustained burns. CACs were isolated and counted under fluorescence microscopy.
Time Frame: baseline
Measure: Mean (Full Range); unit: cells per standard well
Arm/Group | Healthy Volunteers | Burn Volunteer
Number analyzed (Participants) | 10 | 31
cells per standard well | 4,000 [3500 to 4500] | 6,500 [6000 to 7000]

2. Primary Outcome: Mean of Circulating Angiogenic Cells in the Blood of Individuals Who Have Sustained a Burn Injury
Description: as for outcome 1
Time Frame: 0 to 24 hours post-operative
Population: Data was only collected for the experimental arm for this outcome measure to assess the change in amount of CACs after burn injury as time progressed.
Measure: Mean (Full Range); unit: cells per standard well
Arm/Group | Healthy Volunteers | Burn Volunteer
Number analyzed (Participants) | 0 | 31
cells per standard well |  | 6500 [6000 to 7000]

3. Primary Outcome: Mean of Circulating Angiogenic Cells in the Blood of Individuals Who Have Sustained a Burn Injury
Description: as for outcome 1
Time Frame: 49 to 72 hours post-operative
Population: Data only collected for the experimental arm for this outcome measure to assess the change in amount of CACs after burn injury as time progressed.
Measure: Mean (Full Range); unit: cells per standard well
Arm/Group | Healthy Volunteers | Burn Volunteer
Number analyzed (Participants) | 0 | 31
cells per standard well |  | 5000 [4000 to 6000]

4. Primary Outcome: Mean of Circulating Angiogenic Cells in the Blood of Individuals Who Have Sustained a Burn Injury
Description: as for outcome 1
Time Frame: 73 hours to 6 weeks post-operative
Population: as for outcome 2
Measure: Mean (Full Range); unit: cells per standard well
Arm/Group | Healthy Volunteers | Burn Volunteer
Number analyzed (Participants) | 0 | 31
cells per standard well |  | 3500 [3000 to 4000]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Healthy Volunteers | Burn Volunteer
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/31
Other Adverse Events (participants affected / at risk) | 0/10 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes